CLINICAL TRIAL: NCT00637182
Title: An OptioExtension of Trial 1033US/0006 to Assess Safety, Tolerability, Efficacy of Anastrozole (ZD1033, Arimidex™) in Treatment of Gynecomastia in Pubertal Boys Given Placebo and to Conduct a Long-Term Safety Follow-Up of Non-Responding Subjects Given Anastrozole in the Previous Trial
Brief Title: Gynecomastia Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Francisco Sapunar - Medical Science Director, Arimidex
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1033US/0016; D5394L00016
Record Dates: First submitted 2008-03-07; First posted 2008-03-17 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Gynecomastia
Keywords: Gynecomastia; Anastrazole; Arimidex; Pubertal; males; boys
MeSH Terms: conditions — Gynecomastia | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anastrozole
  Other Names: ZD1033; Arimidex™

SUMMARY:
The purpose of this study is to look at the effect of anastrozole (ZD1033, Arimidex™) in reducing gynecomastia in pubertal boys treated with placebo in Trial 1033US/0006 (another anastrozole study).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have entered Trial 1033US/0006 and completed 6 months of treatment and one month of follow-up.
* Subjects must have gynecomastia, with one breast measuring at least 3 cm in diameter.

Exclusion Criteria:

* Subjects who have been given medications known to cause gynecomastia within the previous 3 months

Ages: 11 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2001-01; Primary Completion 2002-06 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Change in linear dimensions of the breast

SECONDARY OUTCOMES:
Change in breast tenderness

CONTACTS AND LOCATIONS:
Overall Officials: Edward O Reiter, MD, Principal Investigator — Baystate Medical Center-Children's Hospital